CLINICAL TRIAL: NCT05750238
Title: Relationship Between Stress, Anxiety, Depression, Sexual Function and Marital Adjustment in Nurses
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Nülüfer Erbil, Prof. Dr., Ordu University
Other Study IDs: september 3
Record Dates: First submitted 2023-01-30; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Stress; Anxiety Disorders; Sexual Behavior
MeSH Terms: conditions — Anxiety Disorders; Sexual Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention, survey was applied to the participants

SUMMARY:
One of the factors that increase harmony in marriage is sexual life and sexual satisfaction (Erdinç, 2018). Sexual intercourse is one of the pillars of a successful family; accordingly, functionality in this area greatly affects marital adjustment (Atrian, 2018). Studies show an important relationship between sexual adjustment and marital adjustment (Türkseven et al., 2020; Begdeş, 2021). Negative workplace factors such as occupational stress and long working hours affect the physical and mental states of nurses (Oyeleye et al., 2013; Chesak et al., 2019).

This study was planned to determine the relationship between stress, anxiety, depression, sexual function and marital adjustment in nurses.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Over the age of 18,
* Married,
* Those whose spouse is alive and living with their spouse will be included.

Exclusion Criteria:

* Having a chronic disease (hypertension, diabetes),
* Nurses who are pregnant,
* Those who use drugs that may affect sexual function (beta-blockers, antihypertensives, antidepressants, antipsychotics, etc.) will be excluded from the study.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — female employees working in the nursing profession were included.
Study Population: female employees working in the nursing profession were included.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Marriage Adjustment Scale Marriage Adjustment Scale | 3 hours
  It is a 15-item Likert-type scale developed by Locke and Wallace (1959) to evaluate marital satisfaction and marital adjustment level. It was adapted into Turkish by Tutarel and Kışlak (1999). The cut-off point of the scale is 43.5. The lowest score obtained from the scale indicates that the woman is very unhappy in her marriage, and the highest score indicates that the woman is very satisfied and happy in her marriage. The Cronbach alpha reliability coefficient in the form of the scale is 0.84 (Tutarel Kışlak, 1999).
Arizona Sexual Experiences Scale | 1 hour
  The Arizona Sexual Experiences Scale (ACEX) was developed by McGahuey et al. (2000) to measure sexual dysfunctions. The scale was adapted to Turkish by Soykan (2004) and its validity and reliability study was conducted. The Women's Form (ACYÖ) Scale is 6-point Likert type and consists of 5 questions. This scale is a Likert-type scale designed to evaluate the five basic components of sexual function: arousal, arousal, vaginal wetting, ability to reach orgasm, and satisfaction with orgasm. Scoring is done from 1 to 6.
Depression, Anxiety and Stress 21 Scale (DASS-21) | 3 hour
  Depression Anxiety Stress-21 Scale (DASS-21); It was developed by Lovibond and Lovibond (Lovibond and Lovibond, 1995) and adapted into Turkish by Sarıçam (Sarıçam, 2017). The scale is likert type and consists of 21 items. There are 7 items in each of the anxiety, depression and stress sub-dimensions. Scale items are scored between "0" and "3", ranging from never to always. The scale evaluates the symptoms of depression, anxiety and stress in the last week. The cut-off score was ≥10 in depression, ≥8 in anxiety, and ≥15 in the stress dimension (Lovibond & Lovibond, 1995). Cronbach alpha internal consistency reliability coefficient of the scale; It was found to be 0.81 for the stress subscale, 0.85 for the anxiety subscale, and 0.87 for the depression subscale (Sarıçam, 2018)

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided